CLINICAL TRIAL: NCT06179628
Title: Low Versus Standard Concentrations and Volumes Local Anesthetics Boluses for Continuous Adductor Canal Block Under Ultrasound-guidance in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Low vs Standard Local Anesthetics Boluses for Continuous Adductor Canal Block in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wirinaree Kampitak, MD, Clinical Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0675/66
Record Dates: First submitted 2023-11-26; First posted 2023-12-22 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Knee Arthropathy
Keywords: Adductor canal block; local infiltration analgesia; Postoperative pain management; Quadriceps strength; Total knee arthroplasty; Local anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Concentration and Volume (Active Comparator): 0.15% bupivacaine 10 ml boluses for continuous adductor canal block
  Interventions: Drug: Low bolus concentration and volume
- Standard Concentration and Volume (Placebo Comparator): 0.25% bupivacaine 20 ml boluses for continuous adductor canal block
  Interventions: Drug: Low bolus concentration and volume

INTERVENTIONS:
Drug: Low bolus concentration and volume — Compare Low and Standard concentrations and volumes of bupivacaine boluses for continuous adductor block
  Other Names: Low concentration and volume of bupivacaine bolus

SUMMARY:
To investigate the efficacy of two different regimens of local anesthetic boluses for continuous adductor canal block under ultrasound-guidance in total knee arthroplasty at King Chulalongkorn Memorial Hospital.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a commonly performed surgical procedure for patients with severe knee osteoarthritis. However, one of the challenges associated with TKA is the significant postoperative pain experienced by patients, which can delay early mobilization and physical therapy. Uncontrolled pain worsens patient outcomes and healthcare costs as it can increase the risk of complications after surgery. Therefore, effective pain management is important for optimizing patient outcomes and promoting a smooth recovery process.Despite the absence of a standardized recommendation for the volume and concentration of bolus administration in continuous adductor canal block (CACB), many previous studies, have demonstrated the efficacy of a high-dose bolus followed by a low-concentration local anesthetic infusion for CACB. However, these trials exhibited differences in the doses and volumes of bolus injection. Therefore, the necessity of high concentration and volume bolus CACB in combination with comprehensive multimodal analgesia and LIA for postoperative pain management in TKA remains uncertain. The aim of this study is to investigate the efficacy of two different regimens of local anesthetic used in boluses for continuous adductor canal block under ultrasound-guidance in total knee arthroplasty at King Chulalongkorn Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TKA aged more than 18 years
* Patients with American Society of Anesthesiologists (ASA) class 1-3
* Patients with body weight index (BMI) 18-40 kg/m2

Exclusion Criteria

* Patient refusal to participate
* Patients with known allergic to medications used in the research protocol
* Patients with contraindications to neuraxial or regional anesthesia, including existing neuropathy or neurological deficits involving the lower extremities, coagulopathy or bleeding diathesis and local skin infections
* Patients with contraindications to NSAIDs such as history of coronary artery bypass graft surgery, congestive heart failure, stroke, gastrointestinal bleedings or ulceration, asthma, hepatic and renal disease, abnormal coagulation, or pregnancy
* Patients with chronic opioid use (opioids have been used daily or almost daily for more than three months or sixty milligrams or more of morphine has been used daily for more than one month) or diagnosed with neuropathic pain
* Patients that are unable to perform preoperative Quantitative sensory testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-12-09 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Average knee pain score assessed by Numerical rating scale (NRS) | 6 hours after surgery
  Average postoperative pain score assessed by NRS from 0-10 (0= no pain, 10= the worst pain imaginable)
Average knee pain score assessed by Numerical rating scale (NRS) | 12 hours after surgery
  Average postoperative pain score assessed by NRS from 0-10 (0= no pain, 10= the worst pain imaginable)

SECONDARY OUTCOMES:
The degree of active range of motion (ROM) of knee joint | preoperative - postoperative day 2
  Evaluate patient's functional outcomes by the degree of knee active ROM (measured by a goniometer) at preoperative and postoperative day 0,1,2
Functional outcomes assessed by Five Times Sit to Stand Test (5XSST) | preoperative - postoperative day 2
  Evaluate patient's functional outcomes by 5XSST at preoperative and postoperative day 0,1,2
Functional outcomes assessed by Time Up and Go (TUG) test | preoperative - postoperative day 2
  Evaluate patient's functional outcomes by TUG tests at preoperative and postoperative day 0,1,2
Postoperative pain score assessed by Numerical rating scale (NRS) | preoperative to day 7 after hospital discharge
  Postoperative pain score at rest and on movement assessed by NRS from 0-10 (0= no pain, 10= the worst pain imaginable)
Quadriceps strength assessed by maximum voluntary isometric contraction (MVIC) in Newton | preoperative - postoperative day 2
  Quadriceps strength assessed by MVIC in Newton at 90 degrees at preoperative and postoperative day 0,1,2
morphine consumption in milligrams | post0perative day 0-2
  Patient's morphine consumption at postoperative day 0,1,2
postoperative complications assessed by Likert scale | postoperative day 0-2
  postoperative complications such as nausea/vomitting, sleep disturbance and fall assessed by Likert scale from 1-7 (1 = strongly disagree/ extremely unlikely, 2 = disagree/ unlikely, 3 = slightly disagree/ slightly unlikely, 4 = either, 5 = slightly agree/ slightly likely, 6 = agree/ likely, 7 = strongly agree/ extremely likely)
The time to first rescue analgesia | postoperative day 0-2
  the period from the CACB administration to the first IV morphine administration

OTHER OUTCOMES:
Length of hospital stay assessed by hours | postoperative day 2
  Evaluate length of hospital stay (from admission to hospital discharge) by hours
patient satisfaction assessed by Numerical rating scale (NRS) | 48 hours after surgery and 7 days after hospital discharge
  Evaluate patient satisfaction by NRS from 0-10 (0= no pain, 10= the worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chadha M, Si S, Bhatt D, Krishnan S, Kumar R, Bansal A, Sharma AK. The Comparison of Two Different Volumes of 0.5% Ropivacaine in Ultrasound-Guided Supraclavicular Brachial Plexus Block Onset and Duration of Analgesia for Upper Limb Surgery: A Randomized Controlled Study. Anesth Essays Res. 2020 Jan-Mar;14(1):87-91. doi: 10.4103/aer.AER_4_20. Epub 2020 Mar 16. PMID 32843799
- [Result] Jaeger P, Jenstrup MT, Lund J, Siersma V, Brondum V, Hilsted KL, Dahl JB. Optimal volume of local anaesthetic for adductor canal block: using the continual reassessment method to estimate ED95. Br J Anaesth. 2015 Dec;115(6):920-6. doi: 10.1093/bja/aev362. PMID 26582853
- [Result] Tao Y, Zheng SQ, Xu T, Wang G, Wang Y, Wu AS, Yue Y. Median effective volume of ropivacaine 0.5% for ultrasound-guided adductor canal block. J Int Med Res. 2018 Oct;46(10):4207-4213. doi: 10.1177/0300060518791685. Epub 2018 Aug 20. PMID 30124351
- [Derived] Kampitak W, Tanavalee A, Ngarmukos S, Wanasrisant N, Homsuwan W. Comparison of 10 mL 0.15% vs 20 mL 0.25% bupivacaine boluses for continuous adductor canal block in total knee arthroplasty: a randomized non-inferiority trial. Reg Anesth Pain Med. 2025 May 20:rapm-2025-106587. doi: 10.1136/rapm-2025-106587. Online ahead of print. PMID 40393775